CLINICAL TRIAL: NCT02594865
Title: Glucerna in Critically Ill Patients (GluCip Trial): Investigating the Glycaemic Effects of a Reduced-carbohydrate, Modified-fat, Fiber-containing Enteral Formula (Glucerna®) in Critically Ill Patients.
Brief Title: The Glycaemic Effects of Glucerna® in Critically Ill Patients.
Acronym: GluCip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PHJ van der Voort (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor-Investigator, PHJ van der Voort, Prof., MD, PhD, MSc, Onze Lieve Vrouwe Gasthuis
Organization: Onze Lieve Vrouwe Gasthuis (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL51918.100.14
Record Dates: First submitted 2015-09-16; First posted 2015-11-03 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Disorder of Glucose Regulation
Keywords: Enteral Nutrition; Continuous Glucose Monitoring
MeSH Terms: interventions — Glucerna; Fresubin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucerna (Active Comparator): Glucerna ® 1.5 kcal (Abbott, USA), the standard enteral formula used at our ICU and the investigational enteral feeding.
  Interventions: Dietary Supplement: Glucerna
- Fresubin (Active Comparator): Fresubin ® Energy Fibre (Fresenius, UK), the control enteral feeding.
  Interventions: Dietary Supplement: Fresubin

INTERVENTIONS:
Dietary Supplement: Glucerna — Glucerna ® 1.5 kcal (Abbott, USA), the standard enteral formula used at our ICU and the investigational enteral feeding.
  Arms: Glucerna
Dietary Supplement: Fresubin — Fresubin ® Energy Fibre (Fresenius, UK), the control enteral feeding.
  Arms: Fresubin

SUMMARY:
To investigate whether the administration of Glucerna achieves less glycaemic variability, defined as the mean absolute glucose (MAG) change, and better glycaemic control compared to a standard high-carbohydrate enteral formula. Continuous glucose monitoring technology will be used to evaluate glycaemic variability and glycaemic control.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patients with an anticipated stay of at least 48 hours of admission to the intensive care
* Expected to receive enteral feeding for at least 48 hrs
* Indication for glucose regulation with insulin (according to the current glucose treatment protocol)
* Patient or surrogate understands and signs informed consent document.

Exclusion Criteria:

* Patients with pre-existing contraindications to enteral feeding or to placement of a continuous glucose monitoring system
* Patients previously randomised into the GluCip trial
* Any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Glucose variability | 72 hours
  The primary outcome is the extent of glucose variability, defined as the mean absolute glucose (MAG) change (delta glucose/delta time) in mmol/l/hr.

SECONDARY OUTCOMES:
Amount of insulin use | 72 hours
  In units/day.
Time in target range | 72 hours
  Defined as a glucose between 6-9 mmol/l in minutes/day.
Mean glucose and standarddeviation | 72 hours
  Defined as the mean sensor glucose and standarddeviation in mmol/l.
Number of severe hypoglycemic events | 72 hours
  Hypoglycemic event is defined as a sensor glucose below 2.2 mmol/l.
Duration of severe hypoglycemic events | 72 hours
  Hypoglycemic event is defined as a sensor glucose below 2.2 mmol/l. Duration is measured in minutes/day.
Number of severe hyperglycemic events | 72 hours
  Hyperglycemic event is defined as a sensor glucose above 15.0 mmol/l.
Duration of severe hyperglycemic events | 72 hours
  Hyperglycemic event is defined as a sensor glucose above 15.0 mmol/l. Duration is measured in minutes/day.
Daily calorie administration | 72 hours
  Defined as amount of calories received per patient/day.
Daily nutrient administration | 72 hours
  Defined as amount of nutrients (carbohydrates, fat, proteins) received per patient/day.

CONTACTS AND LOCATIONS:
Overall Officials: Peter HJ van der Voort, Prof. dr., Principal Investigator — Onze Lieve Vrouwe Gasthuis
Locations (1):
- Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland, Netherlands